CLINICAL TRIAL: NCT01727427
Title: Prospective Study on the Treatment of Unsuspected Pulmonary Embolism in Cancer Patients
Status: Completed | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Marcello Di Nisio, Principal Investigator, G. d'Annunzio University
Other Study IDs: 215/2012
Record Dates: First submitted 2012-11-07; First posted 2012-11-16 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Unsuspected Pulmonary Embolism
Keywords: Unsuspected; pulmonary embolism; cancer
MeSH Terms: conditions — Pulmonary Embolism; Neoplasms | interventions — Heparin; Fondaparinux; Aspirin; Enoxaparin; Dalteparin; Nadroparin; Tinzaparin; bemiparin; Warfarin; Acenocoumarol; Phenprocoumon; Dabigatran; Rivaroxaban; apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Anticoagulants, aspirin: Parenteral or oral anticoagulants: heparin, fondaparinux, vitamin-K antagonists, direct thrombin inhibitors, direct factor Xa inhibitors; aspirin. Any dosage, frequency and duration
  Interventions: Drug: Heparin, fondaparinux, vitamin-K antagonists, aspirin

INTERVENTIONS:
Drug: Heparin, fondaparinux, vitamin-K antagonists, aspirin — Parenteral or oral anticoagulant Antiplatelet agent
  Other Names: Enoxaparin (Clexane); Dalteparin (Fragmin); Nadroparin (Fraxiparin); Tinzaparin (Innohep); Bemiparin (Ivor); Fondaparinux (Arixtra); Warfarin (Coumadin); Acenocoumarol (Sintrom); Phenprocoumon (Marcoumar); Acetylsalicylic acid (Aspirin); Dabigatran (Pradaxa); Rivaroxaban (Xarelto); Apixaban (Eliquis)

SUMMARY:
The same initial and long-term anticoagulation is suggested for unsuspected pulmonary embolism as for patients with symptomatic embolism. Based on these indications, cancer patients with unsuspected pulmonary embolism would be anticoagulated for at least 6 months or until the disease is active, which in most cases would mean indefinite treatment. In fact, dedicated studies on the treatment of unsuspected pulmonary embolism are missing, leaving doubts over the need for (indefinite) anticoagulation which exposes these patients to an increased risk of major bleeding events. Concerns over the need for anticoagulant treatment may especially hold for pulmonary embolism of the distal pulmonary tree since segmental and sub-segmental PE seem to have a more benign course than more proximal embolism.

The scope of this study is to evaluate the current treatment approaches for unsuspected pulmonary embolism and to assess their efficacy and safety in a large prospective cohort of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients with a first diagnosis of unsuspected PE

Exclusion Criteria:

1. age <18 years;
2. ongoing anticoagulant therapy for previous VTE or indications for long-term anticoagulation other than deep vein thrombosis (DVT) or PE;
3. life expectancy less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ambulatory or hospitalized cancer patients with a first diagnosis of unsuspected PE. Both solid and hematological cancers at any stage of disease will be considered for inclusion
Sampling Method: Probability Sample
Enrollment: 695 (Actual)
Dates: Start 2012-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Recurrent (symptomatic) vein thromboembolism, including pulmonary embolism and deep vein thrombosis | one year
  Suspected recurrent PE with one of the following:
  1. new intra-luminal filling defect on CT scan, MRI scan, or pulmonary angiogram;
  2. new perfusion defect of at least 75% on V/Q lung scan;
  3. inconclusive spiral CT, pulmonary angiography or lung scan with demonstration of DVT in the lower extremities by CUS or venography
  Fatal PE is:
  1. PE based on objective diagnostic testing or autopsy or
  2. death not attributed to a documented cause and for which DVT/PE cannot be ruled out.
  Suspected (recurrent) DVT with one of the following findings:
  1. abnormal CUS;
  2. an intra-luminal filling defect on venography.

SECONDARY OUTCOMES:
Major, clinically relevant non-major bleeding, and minor bleeding | one year
  Major bleeding will be defined as overt bleeding associated with: a fall in hemoglobin of 2 g/dL or more, or leading to a transfusion of 2 or more units of packed red blood cells or whole blood, or bleeding that occurs in a critical site: intracranial, intra-spinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal or contributing to death.
  Other clinically relevant non-major bleeding will be defined as overt bleeding not meeting the criteria for major bleeding but associated with medical intervention, unscheduled contact (visit or telephone call) with a physician, (temporary) cessation of study treatment, or associated with discomfort for the patient such as pain, or impairment of activities of daily life. All other bleeding events will be classified as minor.

OTHER OUTCOMES:
Mortality | one year
  Overall mortality

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Di Nisio, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (46):
- D.C. Veterans Affairs Medical Center, Washington D.C., District of Columbia, United States
- Clinical Division of Haematology, Department of Medicine I, Vienna, Austria
- Division of Hematology, University of Ottawa, Ottawa, Canada
- France (15):
  - CHU Amiens Picardie, Amiens
  - Arras/Onco Nord Pas de Callais, Loos, Arras
  - Hopital Saint André, Bordeaux
  - Brest HIA Clermont Tonnerre, Brest
  - University hospital Centra La Cavale Blanche, Brest
  - Montpellier et clinique du parc a Castelnau le nez, Castelnau
  - Hopital G. Montpied Clermont-Ferrand, Clermont
  - AP-HP Hopital Louis Mourier, Colombes
  - Laboratoire d'Hématologie, Dijon, Dijon
  - CHU de Limoges, Limoges
  - Centre Hospitalier Lyon-Sud, Lyon
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Loriboisière, Paris
  - Hospital Pitie Salpetriere, Paris
  - Service de médecine et Thérapeutique, Saint-Etienne
- Division of Vascular Medicine, Department of Medicine, Technical University Dresden, Dresden, Germany
- Italy (6):
  - Ospedali Riuniti, Bergamo
  - Universita degli Studi G. d'Annunzio Chieti e Pescara, Chieti
  - Malattie Cardiovascolari e Nefrourologiche, Palermo
  - Fondazione IRCCS, Pavia
  - Azienda Ospedaliera Arcispedale Santa Maria Nuova (ASMN), Reggio Emilia
  - Università dell'Insubria, Varese
- Netherlands (3):
  - Slotervaart hospital, Amsterdam
  - Academic Medical Center, Amsterdam
  - National Cancer Institute - Antonie van Leeuwenhoek hospital, Amsterdam
- Spain (18):
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de Sabadell, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - ICO_Hospital Duran i Reynals, Barcelona
  - Hospital Clinico Benidorm, Alicante, Benidorm
  - Hospital Universitario Insular de Gran Canarias, Las Palmas
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario de Móstoles, Madrid
  - Hospital Universitario Infantia Sofia, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario San Carlos, Madrid
  - Hospital Santa María Nei, Ourense
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Obispo Polanco, Teruel
  - Hospital Nuestra Sra del Prado Talavera de la Reina, Toledo
  - Hospital Universitario Dr. Peset, Valencia

REFERENCES:
- [Derived] Kraaijpoel N, Bleker SM, Meyer G, Mahe I, Munoz A, Bertoletti L, Bartels-Rutten A, Beyer-Westendorf J, Porreca E, Boulon C, van Es N, Iosub DI, Couturaud F, Biosca M, Lerede T, Lacroix P, Maraveyas A, Aggarwal A, Girard P, Buller HR, Di Nisio M; UPE investigators. Treatment and Long-Term Clinical Outcomes of Incidental Pulmonary Embolism in Patients With Cancer: An International Prospective Cohort Study. J Clin Oncol. 2019 Jul 10;37(20):1713-1720. doi: 10.1200/JCO.18.01977. Epub 2019 May 22. PMID 31116676